CLINICAL TRIAL: NCT03103633
Title: Effects of Perioperative Goal-Directed Therapy Based on Individualized Oxygen Balance on Outcomes During High-risk Cardiac Surgery:A Single Center, Prospective,Randomized,Controlled,Double Blinded Study.
Brief Title: The Effects of Individualized Oxygen Dynamic on Prognosis of Patients With High-risk Cardiac Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The First Affiliated Hospital of Anhui Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: FirstAnhuiM
Record Dates: First submitted 2017-04-01; First posted 2017-04-06 (Actual); Last update posted 2019-03-25 (Actual); Status verified 2017-04

CONDITIONS: Cardiac Disease; High Risk Sex
Keywords: oxygen dynamics; Prognosis
MeSH Terms: conditions — Heart Diseases; Unsafe Sex | interventions — Consciousness Monitors; Control Groups

STUDY DESIGN:
Intervention Model Description: Interventional group:MAP declined with less than 20% of baseline, BIS 45-60 before and after CPB; and BIS 40-45 during CPB, Brain oxygen saturation declined with less than 20% of baseline.
  Control group：no intervention beside the same monitoring with MAP, BIS and brain oxygen saturation and receiving standard measures to achieve a heart rate (HR) in the range of 60-100 beats/min, central venous oxygen saturation (Svco2) higher than 70%, lactate level lower than 3 mmol/L, hematocrit value higher than 28%, and urinary output higher than 0.5 mL/kg/hr.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Patients were followed up by an investigator unaware of the patients' achievement or not of the oxygen dynamic goal
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Individualized Goal-Directed Therapy (Experimental): The goal of intervention:mean artery pressure declined with less than 20% of baseline, BIS 45-60 before and after CPB; and BIS 40-45 during CPB, Brain oxygen saturation declined with less than 20% of baseline.
  Interventions: Procedure: mean artery pressure; Procedure: bispectral index; Procedure: Brain oxygen saturation
- Controlled (Sham Comparator): no intervention beside the same monitoring with MAP, BIS and brain oxygen saturation and receiving standard measures to achieve a heart rate (HR) in the range of 60-100 beats/min, central venous oxygen saturation (Svco2) higher than 70%, lactate level lower than 3 mmol/L, hematocrit value higher than 28%, and urinary output higher than 0.5 mL/kg/hr.
  Interventions: Other: Controlled

INTERVENTIONS:
Procedure: mean artery pressure — mean artery pressure declined with less than 20% of baseline
  Arms: Individualized Goal-Directed Therapy
Procedure: bispectral index — BIS 45-60 before and after CPB; and BIS 40-45 during CPB
  Other Names: BIS
  Arms: Individualized Goal-Directed Therapy
Procedure: Brain oxygen saturation — Brain oxygen saturation declined with less than 20% of baseline
  Arms: Individualized Goal-Directed Therapy
Other: Controlled — receiving standard measures to achieve a heart rate (HR) in the range of 60-100 beats/min, central venous oxygen saturation (Svco2) higher than 70%, lactate level lower than 3 mmol/L, hematocrit value higher than 28%, and urinary output higher than 0.5 mL/kg/hr.
  Arms: Controlled

SUMMARY:
Anesthesia-related factors have been linked to poor perioperative outcomes. Our observational study suggested that the cumulative duration of a triple-low state [intraoperative low mean arterial pressure (MAP), low bispectral index (BIS), and low target effect-site concentration(Ce) ]was associated with poorer 30-day mortality.This randomized, prospective study based on individualized Oxygen dynamics is designed to confirm this association in high-risk patients cardiopulmonary bypass (CPB).

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent;
2. Selective cardiac surgery and general anesthesia patients;
3. Age 18-90 yrs;
4. Anesthesia Society of American (ASA) Scale II-IV
5. European System for Cardiac Operative Risk Evaluation score equal to or greater than 6 or left ventricular ejection fraction lower than 50%

Exclusion Criteria:

1. Preoperative cardiac ejection fraction<30 %;
2. History of anesthesia awareness;
3. History or anticipation of difficult intubation;
4. Unanticipated intraoperative conditions, including haemorrhage, obstinate resuscitation failure,multiple cardiopulmonary bypass procedures, severe hypotension or hypoxemia;
5. long-term preoperative use of anticonvulsant agents, opiates, benzodiazepines or cocaine.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 286 (Actual)
Dates: Start 2017-03-05 (Actual); Primary Completion 2018-06-30 (Actual); Study Completion 2018-07-30 (Actual)

PRIMARY OUTCOMES:
Major postoperative complications(i.e., Rate of low cardiac output syndrome, stroke, myocardial ischemia, infection,reoperation, and need for dialysis) | 30-day after surgery
  Number of Participants with major complications extracted after 30-day follow-up
30-day mortality | 30-day after surgery
  Data for duration of postoperative 30-day all-cause mortality
The change of incidence of postoperative delirium | The 1,2,3 day after surgery
  Through Confusion Assessment Method (CAM)to assess the incidence of the postoperative delirium
1,3,5-year mortality | 1,3,5-year after surgery
  Data for duration of 1,3,5-year all-cause mortality is extracted after 1-year follow-up

SECONDARY OUTCOMES:
postoperative hospital stay | 30-day after surgery
  Data for duration of postoperative hospital stay is extracted after 30-day follow-up
The change of incidence of postoperative cognition dysfunction | 1 day before surgery, the 3,7 day after the surgery
  The neuropsychological tests performed at the day before the surgery,the 3,7 day after the surgery respectively.
The occurrence of cardiovascular events | 30-day after surgery
  Data for duration of the occurrence of cardiovascular events is extracted 30-day follow-up
The incidence of any adverse events | 30-day after surgery
  Including kidney or brain related adverse events 30-day after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Anhui Medical University, Hefei, Anhui, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Cheng XQ, Zhang JY, Wu H, Zuo YM, Tang LL, Zhao Q, Gu EW. Outcomes of individualized goal-directed therapy based on cerebral oxygen balance in high-risk patients undergoing cardiac surgery: A randomized controlled trial. J Clin Anesth. 2020 Dec;67:110032. doi: 10.1016/j.jclinane.2020.110032. Epub 2020 Sep 1. PMID 32889413